CLINICAL TRIAL: NCT06216665
Title: Effect of Pulsatile Hormone Administration on Insulin Action
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Candida Rebello, Assistant Professor, Pennington Biomedical Research Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PBRC 2023-018
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Participants receive insulin delivered continuously or every five minutes during the hyperinsulinemic euglycemic clamp test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous insulin at 40mU/m2/min (Active Comparator): Paricipants will receive insulin infused continuously during the hyperinsulinemic euglycemic clamp test of insulin sensitivity.
  Interventions: Other: Continuous Insulin administration during hyperinsulinemic euglycemic clamp test
- Pulsatile insulin at 40mU/m2/min (Experimental): Participants will receive insulin infused every five minutes during the hyperinsulinemic euglycemic clamp test of insulin sensitivity
  Interventions: Other: Pulsatile Insulin administration during hyperinsulinemic euglycemic clamp test

INTERVENTIONS:
Other: Continuous Insulin administration during hyperinsulinemic euglycemic clamp test — Participants will receive insulin delivered continuously during the hyperinsulinemic euglycemic clamp test
  Arms: Continuous insulin at 40mU/m2/min
Other: Pulsatile Insulin administration during hyperinsulinemic euglycemic clamp test — Participants will receive insulin delivered every five minutes during the hyperinsulinemic euglycemic clamp test
  Arms: Pulsatile insulin at 40mU/m2/min

SUMMARY:
In humans, insulin is secreted in pulses from the pancreatic beta-cells, and these oscillations help to maintain fasting plasma glucose levels within a narrow normal range. Given the fluctuations in insulin concentrations, oscillations enhance precision of control. The hyperinsulinemic euglycemic clamp test (clamp) involves a continuous infusion of insulin and is the gold standard for measuring insulin sensitivity. In this study, insulin sensitivity measured using the standard clamp will be compared with a clamp in which the same total amount of insulin as the standard clamp is infused every five minutes instead of continuously.

DETAILED DESCRIPTION:
Participants with obesity and insulin resistance completing a randomized, controlled, two-arm parallel trial (Motivate) will be enrolled in this cross-sectional study. Twelve participants from the Motivate study will return within two weeks to complete two clamp tests within a week of each other. At these clamps, the insulin will be infused continuously at a dose of 40mU/m2/min during the first clamp test and the same total amount of insulin will be infused every five minutes at the second clamp. The day following the clamps, participants will return to the clinic in a fasted state and blood will be drawn for measurement of glucose and insulin.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the Motivate Study (NCT05649176)

Exclusion Criteria:

* Non-completion of the end-of-study hyperinsulinemic euglycemic clamp test of the Motivate study

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | One day
  Glucose infusion rate during the hyperinsulinemic euglycemic clamp test

SECONDARY OUTCOMES:
Insulin resistance | 24 hours
  Homeostasis Model Assessment of Insulin Resistance

CONTACTS AND LOCATIONS:
Overall Officials: Candida Rebello, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rebello CJ, Morales TS, Chuon K, Dong S, Lam VT, Purner D, Lewis S, Lakey J, Beyl RA, Greenway FL. Physiologic hormone administration improves HbA1C in Native Americans with type 2 diabetes: A retrospective study and review of insulin secretion and action. Obes Rev. 2023 Dec;24(12):e13625. doi: 10.1111/obr.13625. Epub 2023 Aug 14. PMID 37580916